CLINICAL TRIAL: NCT04235894
Title: An Observer Rating Scale of Facial Expression Can Predict Dreaming in Propofol Anesthesia
Status: Completed | Type: Observational
Sponsor: Osijek University Hospital (Other)
Collaborators: Josip Juraj Strossmayer University of Osijek (Other)
Responsible Party: Sponsor
Other Study IDs: Osijek UH
Record Dates: First submitted 2020-01-01; First posted 2020-01-22 (Actual); Last update posted 2020-01-22 (Actual); Status verified 2020-01

CONDITIONS: Anesthesia; Propofol; Drug Effect
Keywords: Propofol;; Endoscopy, Gastrointestinal;; Dreams;; Facial expression;; Smiling
MeSH Terms: conditions — Facial Expression; Smiling | interventions — Propofol

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients undergoing GI endoscopy at Osijek University Hospital: Observational study. A total of 130 consecutive patients undergoing gastrointestinal endoscopy were included. The anesthesia was provided with propofol, starting with 0,5 mg/kg, and titrated until a patient was unresponsive to painful stimuli and maintaining spontaneous breathing. The blood pressure, pulse and Bispectral index values were measured in 6 defined points. On the emergence from anesthesia, the patient's facial expression was rated numerically by the investigator.
  Interventions: Drug: Propofol

INTERVENTIONS:
Drug: Propofol — Intravenous anesthesia with propofol started with 0.5 mg kg-1, and was titrated until a patient was unresponsive to painful stimuli & maintaining spontaneous breathing during gastrointestinal endoscopy
  Other Names: Diprivan

SUMMARY:
This study investigates correlation between dreaming in propofol anesthesia and an Observer-rating-scale of facial expression after gastrointestinal endoscopy in adults. It also compares dreamers and non-dreamers in age, BMI, propofol dose, duration of procedure, mean arterial pressure, pulse values and Bispectral index values.

DETAILED DESCRIPTION:
After Ethical committee approval and written informed consent was obtained, a total of 124 patients undergoing gastrointestinal endoscopy were recruited in the prospective observational study. Anesthesia was maintained using incremental propofol doses until the patient was calm and unresponsive to painful stimuli. Bispectral Index (BIS), blood pressure (BP) and pulse were monitored in typical intervals: before induction, during induction, at the beginning of the procedure, at 2nd, 5th and 10th minute of the procedure, and on emergence. On the emergence of anesthesia, the patient's facial expression was rated numerically (-3 pain, +3 smile). Thereafter patients were asked to rate their dream.

ELIGIBILITY:
Inclusion Criteria:

* Consecutive patients undergoing gastrointestinal endoscopy at Osijek University HOspital form September 2016 to October 2017.

Exclusion Criteria:

* . Patients who were younger than 18 years, unscheduled patients who were not hemodynamically stable, those who were not able to understand study protocol, and who did not sign written informed consent were not included in the study. Patients whose procedure was longer than 60 minutes and patients with incomplete records were excluded from the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive male and female adult patients undergoing gastrointestinal endoscopy at Osijek University Hsspital who wrote informad consent and were able to understand study protocol.
  Patients younger than 18 years, those allergic to propofol and unable to understand study protocol were not included in the study. patients with procedures lasting less than 5 minutes and more than 60 minutes were excluded from the study.
Sampling Method: Non-Probability Sample
Enrollment: 124 (Actual)
Dates: Start 2016-09-07 (Actual); Primary Completion 2017-10-18 (Actual); Study Completion 2017-10-18 (Actual)

PRIMARY OUTCOMES:
Observer rating score after the procedure | On the emergence of anesthesia, max. 2 hours after start of anesthesia
  On the emergence of anesthesia, Observer's: rating of facial expression was written (-3: loud expression of pain; -2: painful grimace; -1: dissatisfaction; 0: neutral; 1: satisfaction; 2: smile and 3: laughter)

SECONDARY OUTCOMES:
Bispectral index values during the procedure | During the propofol anesthesia, max. 2 hours after start of anesthesia
  Bispectral index (BIS) was measured in six points during the procedure; right before the anesthesia, one minute after the first propofol dose, immediately after the start of intervention, 2 minutes after the start of endoscopy, 5 minutes after the start of endoscopy, and finally on the emergence from anesthesia.
Blood pressure values during the procedure | During the propofol anesthesia, max. 2 hours after start of anesthesia
  Blood pressure value was measured in six points during the procedure; right before the anesthesia, one minute after the first propofol dose, immediately after the start of intervention, 2 minutes after the start of endoscopy, 5 minutes after the start of endoscopy, and finally on the emergence from anesthesia.
Pulse values during the procedure | During the propofol anesthesia, max. 2 hours after start of anesthesia
  Pulse value was measured in six points during the procedure; right before the anesthesia, one minute after the first propofol dose, immediately after the start of intervention, 2 minutes after the start of endoscopy, 5 minutes after the start of endoscopy, and finally on the emergence from anesthesia.

CONTACTS AND LOCATIONS:
Overall Officials: Helena Matus, MD, Principal Investigator — Department of emergency medicine, Brodsko-posavska county; Croatia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Leslie K, Kave B. Complications and unplanned admissions in nonoperating room procedures. Curr Opin Anaesthesiol. 2017 Dec;30(6):658-662. doi: 10.1097/ACO.0000000000000519. PMID 28915133
- [Background] Wang D, Chen C, Chen J, Xu Y, Wang L, Zhu Z, Deng D, Chen J, Long A, Tang D, Liu J. The use of propofol as a sedative agent in gastrointestinal endoscopy: a meta-analysis. PLoS One. 2013;8(1):e53311. doi: 10.1371/journal.pone.0053311. Epub 2013 Jan 8. PMID 23308191
- [Background] Koroglu G, Tezcan AH. A Case Report of the First Propofol Addiction in Turkey. Turk J Anaesthesiol Reanim. 2015 Dec;43(6):434-6. doi: 10.5152/TJAR.2015.54872. Epub 2015 Dec 1. PMID 27366543
- [Background] Levy RJ. Clinical effects and lethal and forensic aspects of propofol. J Forensic Sci. 2011 Jan;56 Suppl 1(0 1):S142-7. doi: 10.1111/j.1556-4029.2010.01583.x. Epub 2010 Oct 15. PMID 20950316
- [Background] Ellett ML. Review of propofol and auxiliary medications used for sedation. Gastroenterol Nurs. 2010 Jul-Aug;33(4):284-95; quiz 296-7. doi: 10.1097/SGA.0b013e3181eac371. PMID 20679780
- [Background] Bryson EO, Frost EA. Propofol abuse. Int Anesthesiol Clin. 2011 Winter;49(1):173-80. doi: 10.1097/AIA.0b013e3181f2bcb0. No abstract available. PMID 21239913
- [Background] Horiuchi A, Nakayama Y, Kajiyama M, Kato N, Kamijima T, Ichise Y, Tanaka N. Safety and effectiveness of propofol sedation during and after outpatient colonoscopy. World J Gastroenterol. 2012 Jul 14;18(26):3420-5. doi: 10.3748/wjg.v18.i26.3420. PMID 22807612
- [Background] Tezcan AH, Ornek DH, Ozlu O, Baydar M, Yavuz N, Ozaslan NG, Dilek K, Keske A. Abuse potential assessment of propofol by its subjective effects after sedation. Pak J Med Sci. 2014 Nov-Dec;30(6):1247-52. doi: 10.12669/pjms.306.5811. PMID 25674117
- [Background] Roussin A, Montastruc JL, Lapeyre-Mestre M. Pharmacological and clinical evidences on the potential for abuse and dependence of propofol: a review of the literature. Fundam Clin Pharmacol. 2007 Oct;21(5):459-66. doi: 10.1111/j.1472-8206.2007.00497.x. PMID 17868199
- [Background] Jeon YT. Propofol as a controlled substance: poison or remedy. Korean J Anesthesiol. 2015 Dec;68(6):525-6. doi: 10.4097/kjae.2015.68.6.525. Epub 2015 Nov 25. No abstract available. PMID 26634074
- [Background] Stait ML, Leslie K, Bailey R. Dreaming and recall during sedation for colonoscopy. Anaesth Intensive Care. 2008 Sep;36(5):685-90. doi: 10.1177/0310057X0803600509. PMID 18853587
- [Background] Xu G, Liu X, Sheng Q, Yu F, Wang K. Sex differences in dreaming during short propofol sedation for upper gastrointestinal endoscopy. Neuroreport. 2013 Oct 2;24(14):797-802. doi: 10.1097/WNR.0b013e3283644b66. PMID 23863717
- [Background] Gyulahazi J, Varga K, Igloi E, Redl P, Kormos J, Fulesdi B. The effect of preoperative suggestions on perioperative dreams and dream recalls after administration of different general anesthetic combinations: a randomized trial in maxillofacial surgery. BMC Anesthesiol. 2015 Jan 28;15(1):11. doi: 10.1186/1471-2253-15-11. eCollection 2015. PMID 25685056
- [Background] Bagchi D, Mandal MC, Basu SR. Arousal time from sedation during spinal anaesthesia for elective infraumbilical surgeries: Comparison between propofol and midazolam. Indian J Anaesth. 2014 Jul;58(4):403-9. doi: 10.4103/0019-5049.138972. PMID 25197107
- [Background] Cascella M, Fusco R, Caliendo D, Granata V, Carbone D, Muzio MR, Laurelli G, Greggi S, Falcone F, Forte CA, Cuomo A. Anesthetic dreaming, anesthesia awareness and patient satisfaction after deep sedation with propofol target controlled infusion: A prospective cohort study of patients undergoing day case breast surgery. Oncotarget. 2017 Apr 19;8(45):79248-79256. doi: 10.18632/oncotarget.17238. eCollection 2017 Oct 3. PMID 29108303
- [Background] Eer AS, Padmanabhan U, Leslie K. Propofol dose and incidence of dreaming during sedation. Eur J Anaesthesiol. 2009 Oct;26(10):833-6. doi: 10.1097/EJA.0b013e32832c500c. PMID 19528807
- [Background] Rosenberg RS, Van Hout S. The American Academy of Sleep Medicine Inter-scorer Reliability program: respiratory events. J Clin Sleep Med. 2014 Apr 15;10(4):447-54. doi: 10.5664/jcsm.3630. PMID 24733993
- [Background] Siclari F, Tononi G. Local aspects of sleep and wakefulness. Curr Opin Neurobiol. 2017 Jun;44:222-227. doi: 10.1016/j.conb.2017.05.008. Epub 2017 May 30. PMID 28575720
- [Derived] Matus H, Kvolik S, Rakipovic A, Borzan V. Bispectral Index Monitoring and Observer Rating Scale Correlate with Dreaming during Propofol Anesthesia for Gastrointestinal Endoscopies. Medicina (Kaunas). 2021 Dec 31;58(1):62. doi: 10.3390/medicina58010062. PMID 35056370